CLINICAL TRIAL: NCT03022851
Title: Prospective, Non-randomized, Pilot Study to Assess Safety and Efficacy of a Novel Atrial Flow Regulator (AFR) in Patients With Pulmonary Hypertension
Brief Title: The Prophet Trial -Pilot Study to Assess Safety and Efficacy of a Novel Atrial Flow Regulator (AFR) in Patients With Pulmonary Hypertension
Acronym: AFR-Prophet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Occlutech International AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Occ2016_04; CIV-16-07-016324 (Other: EUDAMED)
Record Dates: First submitted 2017-01-10; First posted 2017-01-18 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2022-09

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Occlutech AFR Device (Experimental): Patients who will get the AFR Device implantation
  Interventions: Device: Occlutech AFR Device

INTERVENTIONS:
Device: Occlutech AFR Device — Catheter-guided transeptal placement of an AFR device following balloon atrial septostomy (BAS) -procedure.

SUMMARY:
This study aims to investigate safety and efficacy of Occlutech® AFR device in patients with severe pulmonary hypertension (PH).

DETAILED DESCRIPTION:
This study will enroll subjects with severe pulmonary hypertension until a maximum of 30 patients have undergone implantation with the Occlutech® AFR device. Enrolment will be devided in 2 phases.

Phase 1: At least 15 adult patients with age ≥ 18 years will be enrolled. Phase 2: Patients with age ≥ 6 years will be enrolled until a maximum of 30 patients is reached.

ELIGIBILITY:
Inclusion Criteria:

1. Age is ≥ 18 / ≥6 years (phase 1 / phase 2).
2. Patient consents to participation
3. The patient or his/her legal representative should have the ability to fluently speak and under-stand the language in which the study is being conducted. If the patient speaks a different language, then a sentence-to-sentence translation for unequivocal understanding must be provided.
4. Written, informed consent by the patient or her/his legally-authorized representative for participation in the study.
5. Patient agrees to comply with the follow-up schedule.
6. Patient has had a successful BAS procedure and is in a stable hemodynamic state, as assessed by the investigator.
7. Conventional treatment options for the patient are exhausted according to ESC and AHA guidelines.
8. SpO2> 86 % pulsoxymetric measurement) This document is confidential and property of Occlutech. It´s only for clinical personnel, Ethical committees and third person in direct contact with the clinical responsible. It is not allowed to distribute information contained in this document without the permission of Occlutech unless the information is already published.
9. "Syncope"(Group A-PH) 9.1. Syncope due to acute PH episodes (as defined by exclusion of other causes) 9.2. Other causes of syncope must have been actively excluded 9.3. Syncope (Black-out) or pre-syncope (episodic dizziness) >2 last 3 months 9.4. PH (defined as mean pulmonary artery pressure > 25 mmHg, or pulmonary vascular resistance of > 3 Wood Units) must exist, RV-failure is however not a prerequisite
10. "RV-Failure"(Group B-PH) 10.1. Right heart failure, chronic and clinically severe 10.1.1.NYHA class III or worse 10.1.2. 6 min walk < 320 m 10.1.3. Signs of venous congestion (distended veins, edema, ascites, etc) 10.1.4.Symptomatic disease resulting in 1 or more PH-related hospitalization over the last 12 months. Elective hospital admissions solely for the purpose of performing diagnostic procedures do not count for this.

10.2. Severe pulmonary hypertension as evident by echocardiography Echocardiographic: 10.2.1. RV larger than LV; 10.2.2. RA larger than LA; 10.2.3. atrial septum bulging into left atrium 10.2.4.ventricular septum bulging into the left ventricle 10.2.5.Reduced (below age-related normal mean value) TAPSE 10.3. Severe pulmonary hypertension as evident by CATH CATH-data: 10.3.1.Mean RA pressure (RAP) of > 10 and ≤ 20 mmHg; 10.3.2.Mean LA pressure (LAP) < 15 mmHg 10.3.3.Mean RAP > mean LAP; 10.3.4.Mean pulmonary arterial pressure >25 mm Hg 10.3.5. Echocardiographically demonstrated continuous right to left shunt following balloon aterial septostomy (BAS) and before AFR device implantation.

Exclusion Criteria

Processes which interfere medically with invasive device implantation

1. Local or generalized sepsis or other acute infection(s)
2. Thrombophilic coagulation disorder
3. Allergy to nickel and/or titanium and/or nickel/titanium-based materials
4. Allergy to anti-platelet, -coagulant, or -thrombotic therapy
5. Intolerance to contrast agents
6. Participation in other medical trials shorter than 30 days before the intended AFR implantation procedure
7. Pregnancy - (assessed in patients with child bearing potential by urine dip stick)
8. Any intracardiac intervention within the last 30 days
9. Thickness of atrial septum > 12mm OR Processes which would technically disturb the safe intervention as planned

1. Occluded inferior vena cava access 2. Previous ASD/PFO closure device in place 3. Intracardiac thrombus OR any other circumstance that, in the opinion of the Investigator,

might interfere with the implantation, might affect the patient's well-being thereafter or might interfere with the conduct and follow up within the Study is general.

Exclusion Criteria:

* Local or generalized sepsis or other acute infection(s)
* Thrombophilic coagulation disorder
* Allergy to nickel and/or titanium and/or nickel/titanium-based materials
* Allergy to anti-platelet, -coagulant, or -thrombotic therapy
* Intolerance to contrast agents
* Participation in other medical trials shorter than 30 days before the intended AFR implantation procedure
* Pregnancy
* Any intracardiac intervention within the last 30 days
* Occluded inferior vena cava access
* Previous ASD/PFO closure device in place
* Intracardiac thrombus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Absence of Serious Adverse Device Effects (SADES) within 3 month following implantation, including deaths, systemic embolism or device embolizations. | 0-3 month
  To evaluate the safety and tolerability of the Occlutech® AFR device by assessing the incidence of SADEs between 3-12 months following implantation.

SECONDARY OUTCOMES:
Rate of all Serious Adverse Events (SAE) and (Serious) Adverse Device Effects (S)ADEs between 3-12 month post implantation | 3-12 month
  To evaluate the safety and tolerability of the Occlutech® AFR device by assessing the incidence of SADEs between 3-12 months following implantation.
Evidence of a secure placement of the device and of right-to-left shunt through the AFR device immediately after implantation and 3 month and 12 month after procedure. | 0-12 month
  The secondary efficacy endpoint will be determined via assessment by color-doppler echocardiography and angiography/fluoroscopy and requires both of:
  Device placed in situ [as assessed by the investigator] Evidence of RIGHT TO LEFT shunt through the AFR device [as assessed by the investigator]
Improvement in number of syncopal events due to pulmonary hypertension in the 3 month, 6 months and 12 month after implantation | 0-12 month

CONTACTS AND LOCATIONS:
Locations (12):
- Germany (3):
  - Klinikum der Universität München, Munich, Bavaria
  - Justus-Liebig Universität, Giesen
  - Universitätsklinikum Würzburg, Würzburg
- Poland (4):
  - Gdański Uniwersytet Medyczny, Gdansk
  - Uniwersytet Jagielloński Collegium Medicum, Krakow
  - Szpital im. Fryderyka Chopina, Otwock
  - Szpital Kliniczny Przemienienia Pańskiego Uniwersytetu Medycznego, Poznan
- Turkey (Türkiye) (5):
  - Hacettepe Üniversitesi Tıp Fakültesi, Ankara, Altındağ
  - Ege Üniversitesi Tıp Fakültesi Hastanesi, Izmir, Bornova
  - Sağlık Bilimleri Üniversitesi Tepecik Eğitim ve Araştırma Hastanesi, Izmir, Konak
  - Ankara Etlik Şehir Hastanesi, Ankara, Yenimahalle
  - Kocaeli Üniversitesi Araştırma ve Uygulama Hastanesi, Kocaeli